CLINICAL TRIAL: NCT00546793
Title: Phase I/II Study of Subcutaneously Administered Veltuzumab (hA20) in Patients With CD20+ Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Brief Title: Ph I/II Study of Subcutaneously Administered Veltuzumab (hA20) in NHL and CLL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hA20-08
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2013-03

CONDITIONS: NHL; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Intermediate-Grade; Lymphoma, Large-Cell; Lymphoma, Low-Grade; Lymphoma, Mixed-Cell; Lymphoma, Small-Cell; Leukemia, Lymphocytic, Chronic; Leukemia, B-Cell, Chronic; Leukemia, Prolymphocytic; Leukemia, Small Lymphocytic; Lymphoma, Small Lymphocytic; Lymphoma, Lymphoplasmacytoid, CLL; Lymphoplasmacytoid Lymphoma, CLL; CLL; SLL
Keywords: humanized anti-CD20 veltuzumab (IMMU-106) administered subcutaneously
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, Follicular; Dendritic Cell Sarcoma, Interdigitating; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Leukemia | interventions — veltuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- veltuzumab (Experimental): veltuzumab is a humanized CD20 antibody administered subcutaneously in this study.
  Interventions: Biological: veltuzumab

INTERVENTIONS:
Biological: veltuzumab — veltuzumab (hA20) will be studied at different dose levels, administered subcutaneously once a week for 4 weeks.
  Other Names: hA20; humanized anti-CD20; IMMU-106

SUMMARY:
The purpose of this study is to determine if a subcutaneous (SC) dosing schedule of veltuzumab can be established in NHL or CLL patients and to confirm the safety and efficacy of veltuzumab that was previously established when administered intravenously.

DETAILED DESCRIPTION:
The first study of veltuzumab given IV weekly in NHL patients (IM-T-hA20-01) has shown excellent tolerability and even efficacy at weekly intravenous doses as low as 80-120 mg/m2 over 4 consecutive weeks. These clinical results confirm experiments laboratory studies. Laboratory studies using Veltuzumab administered subcutaneously showed potent activity based on B-cell depletion. The current study's goal is to determine if a subcutaneous (SC) dosing schedule of veltuzumab can be established in patients with NHL or CLL

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of CD20 positive chronic lymphocytic leukemia (CLL)
* Either previously untreated or relapsed
* Measurable disease (at least one lesion > 1.5 cm for NHL, or ALC > 5,000 for CLL) see full protocol for additional criteria

Exclusion Criteria:

* Previously untreated NHL patients with Stage I and II disease (Ann Arbor classification)
* Previously untreated CLL patients with Stage 0-2 disease (Rai classification) unless specific treatment indications by NCCN guidelines exist (symptomatic, recurrent infections, end-organ function, cytopenias and steady disease progression).

see full protocol for additional criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability | over 2 years after treatment
  safety will be assessed by monitoring lab results and adverse events, which will be assessed every 3 months for up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, PhD, Study Director — Gilead Sciences
Locations (5):
- United States (5):
  - Lewis Cancer Center and Research Pavilion, Savannah, Georgia
  - Cancer Care at Saint Clare's/Saint Clares Hospital Oncology & Hematology Specialists, P.A., Denville, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - New York Hospital Weill Cornell Medical Center, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio

REFERENCES:
- [Background] Morschhauser F, Leonard JP, Coiffier B Petillon M, Coleman M,. Bahkti A, Teoh N, Wegener WA, Goldenberg DM. Phase I/II result of a second-generation humanized anti-CD20 antibody, IMMU-106 (.hA20), in NHL: 2006 ASCO Annual Meeting.Proceedings; 24/18S Part I of II:429s.
- [Background] Morschhauser F, Leonard JP, Fayad L, Coiffier B, Petillon M, Coleman M,. Horne H, Teoh N, Wegener WA, Goldenberg DM. Low doses of humanized anti-CD20 antibody, IMMU-106 (hA20), in refractory or recurrent NHL: Phase I/II results. 2007 ASCO Annual Meeting.Proceedings; 25/18S Part I of II:449s.
- [Background] Stein R, Qu Z, Chen S, Rosario A, Shi V, Hayes M, Horak ID, Hansen HJ, Goldenberg DM. Characterization of a new humanized anti-CD20 monoclonal antibody, IMMU-106, and Its use in combination with the humanized anti-CD22 antibody, epratuzumab, for the therapy of non-Hodgkin's lymphoma. Clin Cancer Res. 2004 Apr 15;10(8):2868-78. doi: 10.1158/1078-0432.ccr-03-0493. PMID 15102696
- [Background] Sapra P, et al. Preclinical pharmacology and toxicology of humanized anti-B-cell antibodies (anti-CD22 and anti-CD20) in cynomolgus monkeys (CM). (Abstract #1471) Blood 2005; 106/11:424a.
- [Background] Stein R, et al. Mechanisms of anti-lymphoma effects of a new humanized anti-CD20 monoclonal antibody, IMMU-106. (Abstract No. 4917) Blood 2003; 102/11:
- [Background] Goldenberg DM, et al. Characterization and preclinical efficacy of hA20, a humanized anti-CD20 monoclonal antibody, for the treatment of NHL. (Abstract #2393) Proceedings of ASCO 2003; 22:595
- [Background] Goldenberg DM, et al. Characterization of new, chimeric and humanized, anti-CD20 monoclonal antibodies, cA20 and hA20, with equivalent efficacy to rituximab in-vitro and in xenografted human non-Hodgkin's lymphoma. (Abstract #2260) Blood 2002; 100/11:575a-576a.
- [Derived] Kalaycio ME, George Negrea O, Allen SL, Rai KR, Abbasi RM, Horne H, Wegener WA, Goldenberg DM. Subcutaneous injections of low doses of humanized anti-CD20 veltuzumab: a phase I study in chronic lymphocytic leukemia. Leuk Lymphoma. 2016;57(4):803-11. doi: 10.3109/10428194.2015.1085531. Epub 2015 Oct 19. PMID 26389849
- [Derived] Negrea GO, Elstrom R, Allen SL, Rai KR, Abbasi RM, Farber CM, Teoh N, Horne H, Wegener WA, Goldenberg DM. Subcutaneous injections of low-dose veltuzumab (humanized anti-CD20 antibody) are safe and active in patients with indolent non-Hodgkin's lymphoma. Haematologica. 2011 Apr;96(4):567-73. doi: 10.3324/haematol.2010.037390. Epub 2010 Dec 20. PMID 21173095